CLINICAL TRIAL: NCT01791998
Title: A Pilot Study to Evaluate Magnet Resonance Thermal Imageguided Interstital Thermal Therapy for Focal Ablation of Breast Cancer
Brief Title: Magnetic Resonance Thermal Image Guided Laser Interstitial Thermal Therapy in Treating Patients With Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was time sensitive and expired. No subjects enrolled.
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1017; NCI-2013-00066 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Ductal Breast Carcinoma in Situ; Invasive Ductal Breast Carcinoma; Stage IA Breast Cancer; Stage IB Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (MR-thermal image guided LITT) (Experimental): Patients undergo MR-thermal image guided LITT over 1 hour.
  Interventions: Procedure: magnetic resonance thermal imaging; Procedure: laser interstitial thermal therapy

INTERVENTIONS:
Procedure: magnetic resonance thermal imaging — Undergo MR-thermal image guided LITT
Procedure: laser interstitial thermal therapy — Undergo MR-thermal image guided LITT

SUMMARY:
This pilot clinical trial studies magnetic resonance thermal image guided laser interstitial thermal therapy in treating patients with breast cancer. Magnetic resonance thermal image guided laser interstitial thermal therapy may be able to kill tumor cells by heating up the tumor cells without affecting the surrounding tissue

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the procedural success rate of using the Visualase magnetic resonance (MR)-guided laser system to target, access, thermally monitor, and focally ablate MR-visible breast cancer lesions.

2. To obtain preliminary data on ablative success using pathologic assessment for specimen excised subsequent to the ablation.

OUTLINE:

Patients undergo MR-thermal image guided laser interstitial thermal therapy (LITT) over 1 hour.

After completion of study treatment, patients are followed up at 3-7 days.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal state
* Histological diagnosis of breast invasive ductal carcinoma with receptor profiles obtained
* MRI visible breast lesion
* Unifocal cancer, less than 1.5 cm in maximum diameter (clinical stage T1), with no evidence of extensive in situ cancer surrounding the main tumor; the eligibility will be determined by the MR imaging appearance of the tumor; if the tumor (proven invasive ductal carcinoma) is a unifocal mass without additional enhancement, it will be judged eligible; however, if the tumor is associated with additional enhancement and/or a satellite focus, it will not judged ineligible, as these are signs of additional in situ or invasive cancer
* Clinical stage N0 (no metastatic axillary lymph node on physical examination or imaging work-up)
* Ability to give informed consent

Exclusion Criteria:

* Previous surgery or radiation for the ipsilateral breast cancer
* Presence of any condition (e.g., metal implant, shrapnel) not compatible with MRI
* Tumor located less than 1 cm from the skin or the pectoralis muscle

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Frequency of not completing the procedure due to patient's discomfort | Up to 7 days
Observed thermal damage on skin | Up to 7 days
  Moderate degree of skin burn which requires medical intervention will be considered side effects for stopping purposes.
Grade 3 or 4 toxicities assessed by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) | Up to 7 days

SECONDARY OUTCOMES:
Amount of tumor necrosis | Up to 7 days
Amount of viable tumor | Up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Abe, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States